CLINICAL TRIAL: NCT03674801
Title: Status of Superficial Esophageal Cancers Treated by Endoscopy
Brief Title: Status of Superficial Esophageal Cancers Treated by Endoscopy "OESOFARE"
Acronym: OESOFARE
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC18_0075
Record Dates: First submitted 2018-07-11; First posted 2018-09-18 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Superficial Esophageal Cancers
Keywords: Superficial esophageal cancer; Endoscopic mucosectomy; Submucosal dissection; therapeutic strategy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In 2013, esophageal cancer was the 9th cause of cancer in the world and the 6th in terms of cancer mortality. The prognosis of this cancer varies according to geographical areas, but in Europe and the USA, the 5-year survival rate has risen from less than 5% in the 1960s to around 20% in the 2000s. In the United States, however, the survival rate has risen from 5% in the 1960s to around 20% in the 2000s.

Increased the detection of premalignant lesions and early stages may improve prognosis. The presence of esophageal cancer is determined by endoscopy, biopsy and histological confirmation. However, endoscopic techniques (mucosectomy and sub mucosal dissection) are also used as curative treatment for early esophageal lesions.

Now, due to the low number of diagnoses of esophageal tumours at the superficial stage, few studies are available in Europe on the efficacy of these endoscopic techniques and on the complications resulting from their use. Similarly, little is known about the complications of endoscopic techniques and about therapeutic strategies for managing these superficial lesions. In particular, no data are available concerning the adequacy between the treatment proposed in multidisciplinary consultation meetings and the actual management of patients.

Our study is therefore fundamental to make an inventory of superficial esophageal cancers treated by endoscopy, and their management

DETAILED DESCRIPTION:
This fundamental study will therefore best describe current French practices for the management strategy of esophageal cancers after endoscopic treatment. Consequently, the interests of this study, national inventory, are multiple:

1. List a significant number of endoscopic treatments. In particular, by sub mucosal dissection in France, in order to strengthen scientific evidence of its efficacy, to assess its feasibility and complication rate.
2. Describe the therapeutic strategies currently in place during endoscopic treatment,
3. Evaluate the adequacy between the proposed upstream management of the endoscopic procedure by SCP and the actual management.

ELIGIBILITY:
Inclusion Criteria:

* Male or female over 18 years of age
* Patient with histologically proven high-grade esophageal cancer (adenocarcinoma or squamous cell carcinoma) or dysplasia
* Patient with digestive endoscopy for endoscopic resection (mucosectomy or submucosal dissection) of a cancerous lesion (adenocarcinoma or squamous cell carcinoma) of the esophagus or high-grade dysplasia.
* Patient who received the study briefing note and agreed to participate

Exclusion Criteria:

* Failure to perform the endoscopic procedure
* Patient under guardianship or guardianship or under judicial safeguard measure
* Pregnant woman
* Patient with prior treatment for esophageal cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The investigator will propose the study to any patient with esophageal cancer (adenocarcinoma or squamous cell carcinoma) or histologically proven high grade dysplasia and having an endoscopy for endoscopic resection of his oesophageal cancer or dysplasia. At least 100 patients will be included in the study
Sampling Method: Non-Probability Sample
Enrollment: 151 (Actual)
Dates: Start 2019-02-26 (Actual); Primary Completion 2022-02-26 (Actual); Study Completion 2025-02-26 (Actual)

PRIMARY OUTCOMES:
Percentage of different managements according to the described method : The Paris endoscopic classification of superficial neoplastic lesions: esophagus, stomach, and colon (Gastrointest. Endosc. 58, S3-43 (2003) | at the endoscopic resection procedure
  In this visit we noted the management by type and histological classification of superficial esophageal tumours

SECONDARY OUTCOMES:
Adequacy between the proposed management before the endoscopic procedure and the actual management | at 3, 6, 12, 18, 24, 30, 36, 42, 48, 54, 60 months
  Percentage of adequacy between the proposed management before the endoscopic procedure and the actual management, defined by the respect of the envisaged strategy and timing
Percentage of complete resection R0 after endoscopic treatment | at 3, 6, 12, 18, 24, 30, 36, 42, 48, 54, 60 months
  Percentage of complete resection R0 after endoscopic treatment
Percentage of patients with endoscopic complication per procedure and/or delayed | at 3, 6, 12, 18, 24, 30, 36, 42, 48, 54, 60 months
  Percentage of patients with endoscopic complication per procedure (esophageal perforation, bleeding) and/or delayed (delayed bleeding, esophageal stenosis)
Percentage of patients treated with mucosectomy or submucosal dissection | at 3, 6, 12, 18, 24, 30, 36, 42, 48, 54, 60 months
  Percentage of patients treated with mucosectomy or submucosal dissection
Number of patients having, in the month following the complementary treatment, an adverse effect | at 3, 6, 12, 18, 24, 30, 36, 42, 48, 54, 60 months
  Number of patients having, in the month following the complementary treatment, an adverse effect such as fever, haemorrhage, retrosternal pain, food blockages or weight loss
Number of patients with a recurrence of cancerous lesion at the initial resection site or at a distance, histologically proven | at 3, 6, 12, 18, 24, 30, 36, 42, 48, 54, 60 months
  Number of patients with a recurrence of cancerous lesion at the initial resection site or at a distance, histologically proven, during follow-up consultations at 3, 6, 12, 18, 24, 30, 36, 42, 48, 54, 60 months post treatment.
Number of patients with recurrence having had a simple monitoring (= therapeutic abstention), endoscopic re-treatment, surgery or radiochemotherapy | at 3, 6, 12, 18, 24, 30, 36, 42, 48, 54, 60 months
  Number of patients with recurrence having had a simple monitoring, endoscopic re-treatment, surgery or radiochemotherapy
"Esophageal Symptoms" questionnaire | at 3, 6, 12, 18, 24, 30, 36, 42, 48, 54, 60 months
  Esophageal Symptoms questionnaires will be filled by the physician at each visit
"SF36" questionnaire | at 3, 6, 12, 18, 24, 30, 36, 42, 48, 54, 60 months
  "SF36" questionnaires will be filled by the physician at each visit

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Nantes, Nantes, France

IPD SHARING:
Plan to Share IPD: No